CLINICAL TRIAL: NCT03137628
Title: Study on the Effect of Conventional General Anesthesia and Mechanical Ventilation on Plasma Small Molecule Metabolites in Patients With Colorectal Cancer Resection
Brief Title: Effect of General Anesthesia and Mechanical Ventilation on Plasma Metabolite in Patient With Colorectal Cancer Resection
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XH-17-005
Record Dates: First submitted 2017-04-24; First posted 2017-05-03 (Actual); Last update posted 2017-05-03 (Actual); Status verified 2017-04

CONDITIONS: Metabolomics
Keywords: general anesthesia,mechanical ventilation,colectomy
MeSH Terms: interventions — Colectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma seperated from venous blood via centrifugation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients undergoing colectomy, GA and MV: venous blood samples collected from colorectal cancer patients undergoing selective colectomy with general anesthesia(GA) and mechanical ventilation(MV) before general anethesia and the third hour after
  Interventions: Other: colectomy, GA and MV
- healthy controls: donated venous blood samples from healthy people undergoing physical examination but not general anesthesia or mechanical ventilation.

INTERVENTIONS:
Other: colectomy, GA and MV — general anesthesia protocol: anesthesia induction (midazolam 0.1mg/kg, sufentanil 0.5ug/kg, etomidate 0.3mg/kg, cisatracurium 0.2mg/kg); anesthesia maintenance [sevoflurane 1.5-3%, cisatracurium 0.1mg/kg/h, sufentanil is supplemented during the entire surgical procedure according to patients' anesthetic situation, dexmedetomidine（used conditionally）0.4ug/kg/h].
  mechanical ventilation protocol: tidal volume 6-8 ml/kg, positive end-expiratory pressure 5 cmH2O, oxygen concentration 40%; respiratory rate 10-15/min, inspiratory/expiratory ratio 1:1.5.
  Groups: patients undergoing colectomy, GA and MV

SUMMARY:
As a newly developed subject, metabolomics can detect accurately and quantitatively small molecule metabolites such as proteins, carbohydrates and lipids from plasma, tissue and even single cell, which aims to analyze systemic dynamic change during physiological and pathological processes, and thus reveals certain reactions that whole organism responds to specific stimulation.

Colorectal cancer is one of common gastrointestinal tumors, whose morbidity rate tends to increase in recent years for modern diet and life style, and colectomy serves as one standard treatment for it. Under total stimulation of surgical operation, general anesthesia and mechanical ventilation, a series of stress reactions happen complicatedly to colorectal patients during anesthesia-ventilation process. Without timely recognition and management of adverse reactions, side effects like hypoxemia, hemorrhage, inflammation, and even death will happen intraoperatively or postoperatively.

With different metabolomics methods applied to collect, detect and analyze blood samples, metabolomics provides an innovatory approach to elucidate systemic response during anesthesia-colectomy process with multi-factors included. By analyzing and comparing dramatic alteration of small molecule metabolites in colorectal cancer patients' or healthy controls' plasma in this project, data can reflect the influence of certain disease (colorectal cancer), anesthetics and mechanical ventilation on colorectal patients with colectomy, which is helpful for prevention and treatment of intraoperative and postoperative complications.

DETAILED DESCRIPTION:
Nowadays, more and more attention are paid to system biology and its relative techniques, such as gene sequencing，nuclear magnetic resonance， mass spectrometry and so on. As a newly developed subject, metabolomics can detect accurately and quantitatively small molecule metabolites such as proteins, carbohydrates and lipids from plasma, tissue and even single cell, which aims to analyze systemic dynamic change during physiological and pathological processes, and thus reveals certain reactions that whole organism responds to specific stimulation.

Colorectal cancer is one of common gastrointestinal tumors, whose morbidity rate tends to increase in recent years for modern diet and life style, and colectomy serves as one standard treatment for it. Under total stimulation of surgical operation, general anesthesia and mechanical ventilation, a series of stress reactions happen complicatedly to colorectal patients during anesthesia-ventilation process. Without timely recognition and management of adverse reactions, side effects like hypoxemia, hemorrhage, inflammation, and even death will happen intraoperatively or postoperatively.

With different metabolomics methods applied to collect, detect and analyze blood samples, metabolomics provides an innovatory approach to elucidate systemic response during anesthesia-colectomy process with multi-factors included. By analyzing and comparing dramatic alteration of small molecule metabolites in colorectal cancer patients' or healthy controls' plasma in this project, data can reflect the influence of certain disease (colorectal cancer), anesthetics and mechanical ventilation on colorectal patients with colectomy, which is helpful for prevention and treatment of intraoperative and postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal cancer patients inclusion criteria: undergo elective colectomy with general anesthesia and mechanical ventilation lasting for > 3.5 hours; classified as physical status I to III according to the American Society of Anesthesiologists Physical Status Classification System; Written informed consent is approved.
* Healthy controls inclusion criteria: volunteers with regular physical examination in nearly three years；without chronic disease; without recent infection in three months; Written informed consent is approved.

Exclusion Criteria:

* Distant metastases; hemodilution with massive fluid supply; recent anaesthetics or mechanical ventilation treatment；children；women during pregnancy or lactation; being involved in other clinical subjects.

Ages: 20 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: colorectal cancer patients and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-03-20 (Actual); Primary Completion 2017-05-05 (Estimated); Study Completion 2017-05-15 (Estimated)

PRIMARY OUTCOMES:
metabolomics | Outcome measure will be assessed right after all samples are collected, which is expected to on May 5, 2017, and MHD files containing compound IDs, m/z values and so on will be reported about 10 days later.
  Thaw Frozen plasma, add methanol and shake. Isolate supernatant after centrifugation. Employ Globle LC-Q-TOF-MS profiling to analyze metabolites of plasma via an Agilent-1200 LC system, coupled with an electrospray Ionization source and an Agilent-6520 Q-TOF mass spectrometry. Utilize Agilent's Mass Hunter Qualitative Analysis Software to process the MS spectra for peak detection, and generate a list detected peak intensities with the retention time-m/z data pairs as identiers. Process integrated raw RHPLC-Q-TOF-MS data with Agilent Mass Hunter Qualitative Analysis and Mass Profiler software. Optimize and choose parameters as follows: the range of m/z values from 80 to 100, and peak filters set to centroid height with > 100 counts, and compound filters set the base peak to > 1000 counts. MHD files will be create, containing compound IDs, and further processing will be performed with Mass Profiler software, which aligns mass features across multiple LC-MS data files.

CONTACTS AND LOCATIONS:
Overall Officials: Lai Jiang, chief doctor, Study Chair — Xinhua Hospital affiliated to Medicine school,Shanghai Jiaotong University
Locations (1):
- Department of Anesthesia, Shanghai Xinhua hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided